CLINICAL TRIAL: NCT04572659
Title: Comparing Different Strategies of Psychosocial Intervention in Assisted Reproduction Treatments
Brief Title: Psychosocial Intervention in Assisted Reproduction Treatments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vida Recoletas Sevilla (Other)
Collaborators: IVI Madrid (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PSYCHOSOCIAL_ART
Record Dates: First submitted 2020-09-17; First posted 2020-10-01 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Infertility Primary; Psychosocial Stressor; Anxiety Depression
Keywords: Assisted Reproduction Treatment (ART); Psychology; Psychosocial intervention; Depression; Anxiety; Life quality
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group intervention (Experimental)
  Interventions: Other: Group psychosocial intervention
- Couple intervention (Experimental)
  Interventions: Other: Couple psychosocial intervention
- No intervention (No Intervention)

INTERVENTIONS:
Other: Group psychosocial intervention — Several couples attended a total of six group psychotherapy sessions conducted by a psychologist. Between 4 and 7 couples were treated in each group session.
  Arms: Group intervention
Other: Couple psychosocial intervention — The couple attended a total of six psychotherapy sessions conducted by a psychologist. Each couple was attended particularly.
  Arms: Couple intervention

SUMMARY:
The aim of the study was to evaluate and compare different strategies of psychosocial intervention for patients undergoing IVF treatment in a private fertility clinic. Recruited patients were assigned to one of three groups: group intervention, couple intervention or no intervention (control group). Three main variables were assessed: depression, anxiety and life quality.

DETAILED DESCRIPTION:
A total of 87 couples have participated in this study. All couples were about to start an assisted reproduction treatment (artificial insemination or in vitro fertilization). Couples were assigned to one of three study groups: group intervention, couple intervention or no intervention (control group). Patients in the first group (group intervention) attended six group psychotherapy sessions. Patients in the second group attended six psychotherapy sessions (particular sessions in this case). The patients in the third group received no psycho-social intervention. Assignation to each group was not randomized, it depended on scheduling availability of the patients. Patients attended one session every week or 15 days. Each session lasted 90 minutes. Sessions were designed to minimize the possible negative psycho -social impact of infertility and its treatment. Different aspects were approached in these sessions including emotion expression, social coping, communication skills, emotion management in different social situations, identification of dysfunctional thoughts, cognitive restructuring, and cognitive distortions. The outcomes measured were: anxiety, depression, life quality, coping and perceived social support. These variables were assessed before ART, after ART and in a follow-up performed six months after ART. Psychological variables were assessed using different well-recognized inventories.

ELIGIBILITY:
Inclusion Criteria:

* Childless couples
* About to undergo an ART treatment

Exclusion Criteria:

* Undergoing ART treatment when signing the informed consent of the study
* Pregnant when signing the informed consent of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2015-03-25 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Depression | 6 months
  Beck's Depression Inventory (BDI-II) (spanish version). Scale from 1 to 40, where a higher score means a more severe depression
Anxiety | 6 months
  State-Trait Anxiety Inventory (STAI) (spanish version). Has 20 items rated on a 4-point scale. Higher scores indicate greater anxiety
Life quality | 6 months
  Fertility Quality of Life (FertiQoL) scoring (spanish version). FertiQoL consists of 36 items scored according to 5 response categories. The response scale has a range of 0 to 4. Higher scores mean higher quality of life.

SECONDARY OUTCOMES:
Coping | 6 months
  Coping Orientation to Problems Experienced (COPE) inventory. 28 item self-report questionnaire. The scale can determine someone's primary coping styles with scores on the following three subscale: Problem-Focussed Coping, Emotion-Focussed Coping, and Avoidant Coping.
Perceived social support (1) | 6 months
  Multidimensional Scale of Perceived Social Support (MSPSS). 12-item measure of perceived adequacy of social support from three sources: family, friends, & significant other; using a 5-point Likert scale.
Perceived social support (2) | 6 months
  Interpersonal Evaluation List (ISEL). Multi- dimensional inventory measuring perceived social support in 40-items

IPD SHARING:
Plan to Share IPD: No